CLINICAL TRIAL: NCT01273467
Title: A Randomized, Double-Blind, Placebo-Controlled Ascending Single-Dose Study of the Intravenous Infusion of CNTO 0007 in Subjects Who Have Experienced Ischemic Cerebral Infarction
Brief Title: A Safety and Tolerability Study of 42037788 (Referred to as CNTO 0007) Compared With Placebo in Patients Who Have Experienced Ischemic Cerebral Infarction (Also Known as Stroke)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016510; 42037788 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Stroke; Ischemia; Infarction
Keywords: Ischemic Cerebral Infarction; Stroke; CNTO0007; 42037788
MeSH Terms: conditions — Stroke; Ischemia; Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): CNTO 0007 or placebo (Stage A) a single IV infusion of a selected dose of CNTO 0007 or placebo administered IV within 1-5 days (depending on cohort) after stroke (first cohort of patients will receive the lowest dose of CNTO 0007 or placebo and each subsequent group will be administered a higher dose (to be determined)
  Interventions: Drug: CNTO 0007 or placebo (Stage A)
- 002 (Experimental): CNTO 0007 or placebo (Stage B) a single IV infusion of the MTD of CNTO 0007 or placebo administered IV within a specified number of days after stroke
  Interventions: Drug: CNTO 0007 or placebo (Stage B)

INTERVENTIONS:
Drug: CNTO 0007 or placebo (Stage A) — a single IV infusion of a selected dose of CNTO 0007 or placebo administered IV within 1-5 days (depending on cohort) after stroke (first cohort of patients will receive the lowest dose of CNTO 0007 or placebo and each subsequent group will be administered a higher dose (to be determined)
  Arms: 001
Drug: CNTO 0007 or placebo (Stage B) — a single IV infusion of the MTD of CNTO 0007 or placebo administered IV within a specified number of days after stroke
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 42037788 (CNTO 0007) in patients who have suffered a stroke. The study is not designed to establish efficacy, although preliminary explorations will be conducted.

DETAILED DESCRIPTION:
This is a first-in-human (FIH) study of 42037788 (referred to as CNTO 0007), a cell therapy being tested to see if it may be useful in treating patients with ischemic cerebral infarction also known as stroke. Patients will be randomized (assigned by chance) to receive a single dose of CNTO 0007 or placebo (identical in appearance to CNTO 0007 but does not contain cells) by intravenous (IV) infusion (injection directly into a vein). Patients and study staff will not know if patients are assigned CNTO 0007 or the placebo. The study will be conducted in 2 stages (Stage A and Stage B). In Stage A, the highest dose of CNTO 0007 that does not cause unacceptable side effects, referred to as the maximum tolerated dose (MTD) will be determined to and administered to patients in Stage B of the study. In Stage A, 5 (up to 7) cohorts (groups) of 4-8 patients each will be administered a single IV infusion of CNTO 0007 or placebo 1-5 days (depending on cohort) after stroke (the first cohort of patients will receive the lowest dose of CNTO 0007 or placebo and each subsequent cohort will be administered a higher dose of CNTO 0007 or placebo until the MTD is determined). In Stage B, patients will be administered a single IV infusion of the MTD within a specified number of days after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have suffered an ischemic stroke, as defined by the protocol (If a woman, must be postmenopausal, defined as having no menses for the 18 months before study start. Premenopausal, surgically-sterilized women must have a negative serum beta human chorionic gonadotropin pregnancy test at screening before CNTO 0007 or placebo administration)
* Patients must be able to remain as inpatients for at least 3 days post-infusion for intensive safety monitoring
* Patients must receive standard post-stroke care before the infusion begins and after treatment with experimental product, including but not limited to appropriate secondary prevention measure such as blood pressure and cholesterol control and antiplatelet agents, unless contraindicated
* Patient must have no clinical evidence of worsening stroke in the last 24 hours prior to the start of the infusion of study treatment
* Patients must have general medical condition consistent with expected survival for at least 1 year.

Exclusion Criteria:

* Presence or history of any clinically significant disease, medical condition, or treatment intervention as determined by the Investigator
* Need for supplementary oxygen for cardiorespiratory reasons or respirator dependency. If supplementary oxygen is not needed for cardiopulmonary reasons but given on a routine basis, it is not exclusionary
* Presence or history of alcohol or drug abuse as defined by the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) within 1 year before the screening phase.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The number and type of adverse events reported | Up to 90 days following study drug administration
Changes in clinical laboratory test values | Up to 90 days following study drug administration
Changes in vital signs measurements | Up to 90 days following study drug administration
Changes in electrocardiograms | Up to 90 days following study drug administration

SECONDARY OUTCOMES:
Blood concentration of CNTO 0007 | At protocol-specified time points on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Portland, Oregon
  - Houston, Texas